CLINICAL TRIAL: NCT05948761
Title: A Randomized Phase 1b-2a Trial of the Safety and Effectiveness of Intermittent Hypoxia Treatment in Parkinson's Disease
Brief Title: Safety and Effectiveness of Intermittent Hypoxia Treatment in Parkinson's Disease
Acronym: TALISMAN-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114210
Record Dates: First submitted 2023-06-20; First posted 2023-07-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Hypoxic conditioning Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identical mode of administration and identical machinery used to deliver the intervention, only inside of machine is different (same ventilator, no active element in the placebo machine)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Hypoxic generator without active elements, pulsewise ventilation assured to ascertain blinding
  Interventions: Other: Normoxia through hypoxic generator without active elements
- Active intervention (Experimental): FiO2 0.16 for 5 minutes interspersed with 5 minutes normoxia (intermittent hypoxia)
  Interventions: Other: Hypoxia through modified hypoxic generator

INTERVENTIONS:
Other: Hypoxia through modified hypoxic generator — Commercially available hypoxic generator, modified to allow for convenient remote interventions by non-expert participants.
  Arms: Active intervention
Other: Normoxia through hypoxic generator without active elements — Commercially available hypoxic generator, modified to allow for convenient remote interventions by non-expert participants, without active elements.
  Arms: Placebo

SUMMARY:
To explore the safety, feasibility and net symptomatic effects of multiple (3x/week, for 4 weeks) intermittent hypoxia treatment sessions in individuals with PD. Secondary outcomes include exploring induction of relevant neuroprotective pathways as measured in serum.

DETAILED DESCRIPTION:
Intermittent hypoxia therapy is a non-pharmacological intervention used by athletes and individuals with cardiovascular disease, amongst others. The safety and feasibility of (intermittent) hypoxia therapy and its short-term effects on Parkinson's disease (PD) symptoms were assessed in a previous exploratory phase I trial. However, the net effects of multiple hypoxia treatment sessions on PD symptoms are unknown. The results of the previous phase I trial informed the study design of the newly proposed phase 1b-2a safety and efficacy trial.

45 minutes of normobaric intermittent hypoxia (FiO2 0.16 for 5 minutes interspersed with 5 minutes normoxia) will be delivered via a hypoxicator (a device that titrates decreased fractional oxygen from room air) through an oxygen mask in the hospital and subsequently at participants' homes. Interventions will be conducted 3 times a week, for 4 weeks in total.

ELIGIBILITY:
Inclusion criteria

* Informed consent
* Clinical diagnosis of Parkinson's disease by a movement disorder specialized neurologist.
* Hoehn and Yahr staging 1 to and including 3 (indicating mild to moderate PD).

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Individuals with diseases leading to restrictive and obstructive pulmonary diseases, sleep apnea and cardiac output deficits, such as pulmonary fibrosis, COPD, sleep apnea or excessive alcoholic intake, and congestive heart failure respectively
* Individuals with coronary artery disease NYHA classes III and IV
* Arterial blood gas abnormalities at screening procedure
* Individuals with shortness of breath or other airway or breathing-related inconvenience related to lack of dopaminergic medication
* Inability for in-clinic measurements in OFF phase
* Individuals with active deep brain stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Number and nature of adverse events | 2 months
Feasibility questionnaire, overall study success | 1 month
  Higher indicates better score

SECONDARY OUTCOMES:
MDS-UPDRS part II and III | 1 month
  Lower indicates better score
Purdue pegboard test (PPT) | 1 month
  Higher indicates better score
Timed up & Go Test (TUGT) | 1 month
  Lower indicates better score
Exercise tolerance (6-minute walk test, 6MWT) | 1 month
  Higher indicates better score
Accelerometry data for tremor amplitude | 1 month
  Lower indicates better score
Accelerometry data for pronation-supination | 1 month
  Higher indicates better score
Hematocrit | 1 month
  Higher indicates better result
Neurofilament light chain (NfL) | 1 month
  Higher indicates better result
BDNF | 1 month
  Higher indicates better result
Platelet-derived growth factor receptor beta (PDGFRβ) | 1 month
  Higher indicates better result
Clusterin | 1 month
  Higher indicates better result
GFAP | 1 month
  Higher indicates better result
UCH-L1 | 1 month
  Higher indicates better result

OTHER OUTCOMES:
Parkinson's disease Questionnaire-39 (PDQ-39) | 1 month
  Lower indicates better score

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Dpt. of Physiology, Radboud University Medical Center, Nijmegen
  - Radboud University Medical Center, Nijmegen

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared with The Michael J. Fox Foundation for Parkinson's Research (the study funder). This data may be kept for storage at a central repository either hosted by The Michael J. Fox Foundation, its collaborators, or consultants and will be kept indefinitely. Anonymized data will be made publicly available for the intended use of research in Parkinson's disease as well as other biomedical research studies that may not be related to Parkinson's disease.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 1.5 years

REFERENCES:
- [Background] Janssen Daalen JM, Meinders MJ, Giardina F, Roes KCB, Stunnenberg BC, Mathur S, Ainslie PN, Thijssen DHJ, Bloem BR. Multiple N-of-1 trials to investigate hypoxia therapy in Parkinson's disease: study rationale and protocol. BMC Neurol. 2022 Jul 14;22(1):262. doi: 10.1186/s12883-022-02770-7. PMID 35836147
- [Derived] Janssen Daalen JM, Meinders MJ, Mathur S, van Hees HWH, Ainslie PN, Thijssen DHJ, Bloem BR. Randomized controlled trial of intermittent hypoxia in Parkinson's disease: study rationale and protocol. BMC Neurol. 2024 Jun 22;24(1):212. doi: 10.1186/s12883-024-03702-3. PMID 38909201